CLINICAL TRIAL: NCT00479973
Title: The Anti-Diabetic and Cholesterol-Lowering Effects of Cinnamon and Cassia Bark (Cinnamomum Verum and C. Aromaticum) (Cinnamonforce™) - Randomized Placebo-Controlled Clinical Trial
Brief Title: The Anti-Diabetic and Cholesterol-Lowering Effects of Cinnamon and Cassia Bark
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Canadian College of Naturopathic Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dug2006-1
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Type 2 Diabetes; Hypercholesterolemia
Keywords: diabetes; non-insulin dependant diabetes; type 2 diabetes; cinnamon; natural health product; hypercholesterolemia; dyslipidemia; elevated cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cinnamonforce (Active Comparator): Cinnamonforce™ is a proprietary blend of Cinnamomum aromaticum and Cinnamomum verum bark containing 47 mg of hydroethanolic extract (min. 8% total phenolics) and 23 mg supercritical extract (min. 35% cinnamaldehyde) per capsule.
  Interventions: Dietary Supplement: Cinnamonforce
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cinnamonforce — Cinnamonforce™ is a proprietary blend of Cinnamomum aromaticum and Cinnamomum verum bark containing 47 mg of hydroethanolic extract (min. 8% total phenolics) and 23 mg supercritical extract (min. 35% cinnamaldehyde) per capsule.
  2 capsules after the two largest meals of the day
  Other Names: Cinnamonforce by New Chapter
  Arms: Cinnamonforce
Dietary Supplement: Placebo — Placebo. 2 capsules after the two largest meals of the day
  Arms: Placebo

SUMMARY:
Introduction: According to the World Health Organization (WHO), approximately 150 million people worldwide have type 2 diabetes. Common and cassia cinnamon have been reported to have anti-diabetic and lipid-lowering effects.

Objective: To determine if the combination common and cassia cinnamon product Cinnamonforce™ (Cinnamomum verum and C. aromaticum) reduces fasting blood glucose, insulin, glycosylated hemoglobin (HA1C), triglyceride, total cholesterol, HDL cholesterol and LDL cholesterol levels in people with type 2 diabetes.

Methodology: Seventy (70) type 2 diabetic participants will be randomized to receive either 140 mg of Cinnamonforce twice daily or placebo over 12 weeks. Physical and laboratory measurements will be taken at baseline, 2 weeks, 4 weeks, 8 weeks and at the end of the trial, 13 weeks.

Results: The differences in the measurements obtained from the group receiving Cinnamonforce and the placebo group will be analyzed and discussed.

DETAILED DESCRIPTION:
A randomized placebo-controlled clinical trial will be conducted to evaluate the impact of Cinnamonforce™ on different serum markers related to diabetes and lipid management. Cinnamonforce™ is a proprietary blend of Cinnamomum aromaticum and Cinnamomum verum bark containing 47 mg of hydroethanolic extract (min. 8% total phenolics) and 23 mg supercritical extract (min. 35% cinnamaldehyde) per capsule. Based on inclusion and exclusion criteria outlined in 13A, seventy (70) participants will be randomized using a computer-derived random number generator to the treatment group where they will receive Cinnamonforce™ or to the control group where they will receive a placebo. The manufacturer of Cinnamonforce™, New Chapter, will generate the treatment allocations and retain these in sealed opaque envelopes until the end of the trial. Patients, investigators, and statisticians will be blinded until the end of the trial. Participants will be administered 140 mg of Cinnamonforce™ twice daily or placebo of identical size, shape, colour and odour. Patients will be instructed to take two capsules (140 mg) at the end of each of the two largest meals of the day for 3 months. Compliance will be assessed by pill count.Participants will be asked to come in for assessment at predefined time points including: baseline, 2 weeks, 4 weeks, 8 weeks and end point (13 weeks). At each time point, objective and subjective measurements will be obtained.

The primary objective measures will consist of fasting blood glucose, insulin and HA1C. Secondary biochemical measures will include a lipid panel (total cholesterol,triglycerides, HDL and LDL). Other secondary objective measures will consist of blood pressure, weight, body mass index (BMI), waist/hip measurements, patient self-monitoring of blood glucose and homeostasis model assessment of insulin resistance (HOMA-IR) calculations. Liver and kidney toxicity of the intervention will be assessed through serum measurements of a liver panel (AST, ALT, total protein, albumin, alkaline phosphatase, total bilirubin and direct bilirubin), creatinine and blood-urea-nitrogen (BUN). Coagulability effects will be measured (PT, PTT, fibrinogen). Subjective tolerability of the treatment and reported adverse effects will also be included as secondary outcomes. Another secondary outcome will consist of subjective scores from self-reported questionnaires,i.e. Diabetes-39, SF-36.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Aged > 30
* Male or female
* Not taking anti-diabetic or lipid-lowering medication OR on a stable drug regimen for at least 3 months without any planned dosage change by the participants attending physician
* Have fasting blood glucose at or between 8-15 mmol/L
* Not taking any medications or natural health products that may affect serum parameters tested
* Having already been educated in exercise and dietary changes known to improve glucose control

Exclusion Criteria:

* Type 1 diabetics
* Patients taking insulin
* Pregnant or planned pregnancy
* Breastfeeding
* Known allergy to ingredients in Cinnamonforce
* Patients with underlying heart, liver, kidney, endocrine or neurologic disease
* Patients on an unstable hypoglycemic or lipid-lowering drug regime or patients on a drug regimen for less than 3 months, and patients taking medication that may affect serum parameters tested

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-09; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
The primary objective measures will consist of fasting blood glucose, insulin and HA1C. | 3 months

SECONDARY OUTCOMES:
Total-C, TG, HDL, LDL, BP, weight, BMI, waist/hip ratio, self-monitoring blood glucose, HOMA-IR, AST, ALT, total protein, albumin, alk phos, total/direct bilirubin, creatinine, BUN, PT, PTT, fibrinogen, adverse effects, Diabetes-39, SF-36 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rowena Ridout, MD, Principal Investigator — UHN; Jean-Jacques Dugoua, ND PhD(cand), Study Director — University of Toronto; Gideon Koren, MD, Study Director — University Toronto; Tom Einarson, PhD, Study Director — University of Toronto
Locations (2):
- Canada (2):
  - Canadian College of Naturopathic Medicine, Toronto, Ontario
  - UHN - Toronto Western Hospital, Toronto, Ontario